CLINICAL TRIAL: NCT03144622
Title: (4S)-4-(3-[18F]Fluoropropyl)-L-glutamate Radiotracer (FSPG) PET/CT for Imaging xC- Transporter Activity in Cancers
Brief Title: 18F-FSPG PET/CT Imaging in Patients With Cancers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201412135MINC
Record Dates: First submitted 2017-04-26; First posted 2017-05-09 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Pulmonary Cancer; Breast Neoplasms; Abdominal Cancer
Keywords: (4S)-4-(3-[18F]fluoropropyl-)-L-glutamate; 18F-FSPG; PET/CT; system xC-transporter
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to compare the diagnostic performance of 18F-FDG and 18F-FSPG PET/CT in lung, breast, and abdominal cancers before undergoing therapy. In addition, the role of 18F-FSPG PET/CT in evaluating therapy response and prognosis will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients are given the opportunity to participate in the study if

  1. Age ≥ 20 years old.
  2. Confirmed diagnosis of primary cancer of the following: NSCLC, breast or abdominal cancers
  3. ECOG performance status 0 to 2.
  4. Life expectancy > 3 months.
  5. Consent to perform additional 18F-FSPG and 18F-FDG PET prior to therapy.
  6. Sexually active subjects agree to use condoms and/or their partners of reproductive potential to use a method of effective birth control during imaging period of 2 weeks.

Exclusion Criteria:

* Patients with any of the following conditions will be excluded

  1. Had received previous treatment (excluding neoadjuvant therapy).
  2. Pregnant or lactating women.
  3. Known malignancy in other organs.
  4. Evaluated by primary care physician as unsuitable.
  5. Known hypersensitivity to the study drug.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical diagnosis of NSCLC, breast, and abdominal cancers
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-09-06 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Staging ability of 18F-FSPG PET/CT | 3 years
  Sensitivity, specificity, diagnostic accuracy of 18F-FSPG and 18F-FDG PET/CT will be compared according to patient-based and lesion-based analysis using paired t-test or Krusal-Wallis test.
Ability of 18F-FSPG PET/CT in therapy response evaluation and prognosis prediction | 3 years
  Comparison between 18F-FSPG and 18F-FDG PET/CT will be done using both qualitative and quantitative measures

SECONDARY OUTCOMES:
Uptake of 18F-FSPG | 3 years
  Standardised uptake values (SUV) will be compared between 18F-FSPG and 18F-FDG
Safety of 18F-FSPG PET/CT | 3 years
  Number of reported adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Fang Cheng, MD, Principal Investigator — National Taiwan University Hospital Department of Nuclear Medicine
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No